CLINICAL TRIAL: NCT02495389
Title: Mirabegron and Urinary Urgency Incontinence: The Clinical Response and the Female Urinary Microbiome
Brief Title: Mirabegron and Urinary Urgency Incontinence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, Alan J. Wolfe, Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 207102
Record Dates: First submitted 2015-07-09; First posted 2015-07-13 (Estimated); Results first posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Overactive Bladder
Keywords: Urinary Urgency Incontinence; Mirabegron; Myrbetriq; Betmiga
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron

STUDY DESIGN:
Intervention Model Description: All patients receive mirabegron daily for 12 weeks
Masking Description: There is no masking scheme
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mirabegron (Experimental): Participants received mirabegron (Myrbetriq) daily for 12 weeks
  Interventions: Drug: Mirabegron

INTERVENTIONS:
Drug: Mirabegron — Mirabegron is a medication for the treatment of overactive bladder. It was developed by Astellas Pharma and was approved by the United States Food and Drug Administration (FDA) in July 2012.
  Other Names: Myrbetriq; Betmiga

SUMMARY:
This study is for women diagnosed with urinary urgency incontinence (UUI) or overactive bladder (OAB). Some patients continue to have symptoms even while taking medication for OAB. The purpose of this study is to estimate the number of women who respond to a medication called mirabegron and estimate change in symptom severity over 12 weeks of therapy. A secondary goal is to correlate the female urinary microbiome (FUM) with response to treatment and change in symptom severity over 12 weeks of therapy.

DETAILED DESCRIPTION:
Mirabegron is an FDA-approved medication for urgency incontinence. Evaluation of mirabegron's influence on clinical symptoms may need to take into account the effect of the female urinary microbiome (FUM) on a patient's response to treatment. Compared to asymptomatic patients, several bacterial species are more common in patients with overactive bladder.

Currently, physicians have limited ability to personalize a patient's urinary urgency incontinence treatment and, consequently, the prescribed medication may provide minimal symptom relief. Since the FUM can be assessed prior to treatment, this study proposes to determine if baseline FUM assessment can provide insight into future symptom relief with mirabegron treatment.

ELIGIBILITY:
Inclusion Criteria:

* Bothersome idiopathic (non-neurologic) urgency urinary incontinence (UUI) who recall ≥ 5 urgency predominant urinary incontinence episodes in the prior week (urgency urinary incontinence or mixed urinary incontinence-urgency predominant)
* No contraindications to taking mirabegron
* Patients on current OAB therapy will undergo a two-week drug washout period prior to baseline assessment

Exclusion Criteria:

* Neurologic disease known to affect the lower urinary tract
* Systemic immunologic deficiency
* Current urinary tract infection (UTI) (based on dipstick assessment) or recurrent culture-proven UTIs
* History or current pelvic malignancy or radiation
* Untreated symptomatic pelvic organ prolapse (POP) > POP-Q Stage II
* A contraindication to receiving mirabegron
* Women of childbearing potential who are pregnant or nursing or intend to become pregnant during the study, or who are not practicing a reliable method of contraception
* Must not have taken any antibiotics in the 4 weeks prior to enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-01-28 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Wolfe, PhD, Principal Investigator — Loyola Univerity Medical Center
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Barber MD, Chen Z, Lukacz E, Markland A, Wai C, Brubaker L, Nygaard I, Weidner A, Janz NK, Spino C. Further validation of the short form versions of the Pelvic Floor Distress Inventory (PFDI) and Pelvic Floor Impact Questionnaire (PFIQ). Neurourol Urodyn. 2011 Apr;30(4):541-6. doi: 10.1002/nau.20934. Epub 2011 Feb 22. PMID 21344495
- [Background] Brubaker L, Nager CW, Richter HE, Visco A, Nygaard I, Barber MD, Schaffer J, Meikle S, Wallace D, Shibata N, Wolfe AJ. Urinary bacteria in adult women with urgency urinary incontinence. Int Urogynecol J. 2014 Sep;25(9):1179-84. doi: 10.1007/s00192-013-2325-2. Epub 2014 Feb 11. PMID 24515544
- [Background] Chapple CR, Cardozo L, Nitti VW, Siddiqui E, Michel MC. Mirabegron in overactive bladder: a review of efficacy, safety, and tolerability. Neurourol Urodyn. 2014 Jan;33(1):17-30. doi: 10.1002/nau.22505. Epub 2013 Oct 11. PMID 24127366
- [Background] Chapple CR, Nitti VW, Khullar V, Wyndaele JJ, Herschorn S, van Kerrebroeck P, Blauwet MB, Siddiqui E. Onset of action of the beta3-adrenoceptor agonist, mirabegron, in Phase II and III clinical trials in patients with overactive bladder. World J Urol. 2014 Dec;32(6):1565-72. doi: 10.1007/s00345-014-1244-2. Epub 2014 Jan 24. PMID 24458878
- [Background] Coyne K, Revicki D, Hunt T, Corey R, Stewart W, Bentkover J, Kurth H, Abrams P. Psychometric validation of an overactive bladder symptom and health-related quality of life questionnaire: the OAB-q. Qual Life Res. 2002 Sep;11(6):563-74. doi: 10.1023/a:1016370925601. PMID 12206577
- [Background] Coyne KS, Matza LS, Kopp Z, Abrams P. The validation of the patient perception of bladder condition (PPBC): a single-item global measure for patients with overactive bladder. Eur Urol. 2006 Jun;49(6):1079-86. doi: 10.1016/j.eururo.2006.01.007. Epub 2006 Jan 24. PMID 16460875
- [Background] de Boer TA, Salvatore S, Cardozo L, Chapple C, Kelleher C, van Kerrebroeck P, Kirby MG, Koelbl H, Espuna-Pons M, Milsom I, Tubaro A, Wagg A, Vierhout ME. Pelvic organ prolapse and overactive bladder. Neurourol Urodyn. 2010;29(1):30-9. doi: 10.1002/nau.20858. PMID 20025017
- [Background] Fouts DE, Pieper R, Szpakowski S, Pohl H, Knoblach S, Suh MJ, Huang ST, Ljungberg I, Sprague BM, Lucas SK, Torralba M, Nelson KE, Groah SL. Integrated next-generation sequencing of 16S rDNA and metaproteomics differentiate the healthy urine microbiome from asymptomatic bacteriuria in neuropathic bladder associated with spinal cord injury. J Transl Med. 2012 Aug 28;10:174. doi: 10.1186/1479-5876-10-174. PMID 22929533
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Background] Hilt EE, McKinley K, Pearce MM, Rosenfeld AB, Zilliox MJ, Mueller ER, Brubaker L, Gai X, Wolfe AJ, Schreckenberger PC. Urine is not sterile: use of enhanced urine culture techniques to detect resident bacterial flora in the adult female bladder. J Clin Microbiol. 2014 Mar;52(3):871-6. doi: 10.1128/JCM.02876-13. Epub 2013 Dec 26. PMID 24371246
- [Background] Irwin DE, Kopp ZS, Agatep B, Milsom I, Abrams P. Worldwide prevalence estimates of lower urinary tract symptoms, overactive bladder, urinary incontinence and bladder outlet obstruction. BJU Int. 2011 Oct;108(7):1132-8. doi: 10.1111/j.1464-410X.2010.09993.x. Epub 2011 Jan 13. PMID 21231991
- [Background] Kenton K, Fitzgerald MP, Brubaker L. What is a clinician to do-believe the patient or her urinary diary? J Urol. 2006 Aug;176(2):633-5; discussion 635. doi: 10.1016/j.juro.2006.03.069. PMID 16813908
- [Background] Khasriya R, Sathiananthamoorthy S, Ismail S, Kelsey M, Wilson M, Rohn JL, Malone-Lee J. Spectrum of bacterial colonization associated with urothelial cells from patients with chronic lower urinary tract symptoms. J Clin Microbiol. 2013 Jul;51(7):2054-62. doi: 10.1128/JCM.03314-12. Epub 2013 Apr 17. PMID 23596238
- [Background] Lowenstein L, Rickey L, Kenton K, Fitzgerald MP, Brubaker L, Tulke M, Fordham J, Mueller ER. Reliability and responsiveness of the Urgency Severity and Life Impact Questionnaire (USIQ). Int Urogynecol J. 2012 Feb;23(2):193-6. doi: 10.1007/s00192-011-1531-z. Epub 2011 Aug 18. PMID 21850507
- [Background] Michel MC, Chapple CR. Basic mechanisms of urgency: roles and benefits of pharmacotherapy. World J Urol. 2009 Dec;27(6):705-9. doi: 10.1007/s00345-009-0446-5. PMID 19588154
- [Background] Mostwin JL. Pathophysiology: the varieties of bladder overactivity. Urology. 2002 Nov;60(5 Suppl 1):22-6; discussion 27. doi: 10.1016/s0090-4295(02)01788-0. PMID 12493346
- [Background] Pearce MM, Hilt EE, Rosenfeld AB, Zilliox MJ, Thomas-White K, Fok C, Kliethermes S, Schreckenberger PC, Brubaker L, Gai X, Wolfe AJ. The female urinary microbiome: a comparison of women with and without urgency urinary incontinence. mBio. 2014 Jul 8;5(4):e01283-14. doi: 10.1128/mBio.01283-14. PMID 25006228
- [Background] Sajadi KP, Vasavada SP. Overactive bladder after sling surgery. Curr Urol Rep. 2010 Nov;11(6):366-71. doi: 10.1007/s11934-010-0136-2. PMID 20803179
- [Background] Siddiqui H, Nederbragt AJ, Lagesen K, Jeansson SL, Jakobsen KS. Assessing diversity of the female urine microbiota by high throughput sequencing of 16S rDNA amplicons. BMC Microbiol. 2011 Nov 2;11:244. doi: 10.1186/1471-2180-11-244. PMID 22047020
- [Background] Smith HS, Hughes JP, Hooton TM, Roberts P, Scholes D, Stergachis A, Stapleton A, Stamm WE. Antecedent antimicrobial use increases the risk of uncomplicated cystitis in young women. Clin Infect Dis. 1997 Jul;25(1):63-8. doi: 10.1086/514502. PMID 9243034
- [Background] Tincello DG, Owen RK, Slack MC, Abrams KR. Validation of the Patient Global Impression scales for use in detrusor overactivity: secondary analysis of the RELAX study. BJOG. 2013 Jan;120(2):212-216. doi: 10.1111/1471-0528.12069. Epub 2012 Nov 27. PMID 23189940
- [Background] Wolfe AJ, Toh E, Shibata N, Rong R, Kenton K, Fitzgerald M, Mueller ER, Schreckenberger P, Dong Q, Nelson DE, Brubaker L. Evidence of uncultivated bacteria in the adult female bladder. J Clin Microbiol. 2012 Apr;50(4):1376-83. doi: 10.1128/JCM.05852-11. Epub 2012 Jan 25. PMID 22278835
- [Derived] Halverson T, Mueller ER, Brubaker L, Wolfe AJ. Symptom improvement with mirabegron treatment is associated with urobiome changes in adult women. Int Urogynecol J. 2022 May;33(5):1319-1328. doi: 10.1007/s00192-022-05190-w. Epub 2022 Apr 12. PMID 35412069

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from January 2015 through October 2018 (46 months) from a tertiary care female pelvic medicine and reconstructive surgery practice.
Groups:
- Mirabegron: This arm comprises women who received mirabegron
Period: Overall Study
Arm/Group | Mirabegron
Started | 84
Completed | 44
Not Completed | 40
Not completed — Withdrawal by Subject | 40

BASELINE CHARACTERISTICS:
Arm/Group | Mirabegron
Number analyzed (Participants) | 84
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One participant did not report her age
  years
    number analyzed (Participants) | 83
    (all) | 66.67 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian or White | 65
  Race: African American or Black | 11
  Race: Asian | 1
  Race: Multiracial | 1
  Race: Other | 4
  Race: Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 84
Hormone Replacement Therapy [Count of Participants; unit: Participants]
  Taking hormone replacement therapy | 7
  Not taking hormone replacement therapy | 75
  Unknown | 2
Type II Diabetes Status [Count of Participants; unit: Participants]
  Diabetic | 16
  Non-Diabetic | 67
  Not reported | 1
Smoker Status [Count of Participants; unit: Participants]
  Smoker | 8
  Non-smoker | 74
  Not reported | 2
Hypertension Status [Count of Participants; unit: Participants]
  Hypertensive | 43
  Non-hypertensive | 40
  Not reported | 1
Cardiovascular Status [Count of Participants; unit: Participants]
  Heart disease | 12
  No heart disease | 71
  Not reported | 1
Chronic Obstructive Pulmonary Disease (COPD) [Count of Participants; unit: Participants]
  Positive | 4
  Negative | 78
  Not reported | 2
Asthma Status [Count of Participants; unit: Participants]
  Positive | 13
  Negative | 69
  Not reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Response to Therapy
Description: Response to therapy was measured using the Patient Perception of Bladder Control (PPBC) questionnaire which measures patients' perceived bladder condition on a 6-point ordinal scale ranging from 1 (no problems at all) to 6 (many severe problems). Women reporting a PPBC score of 4 or 5 by week 12 responded to therapy. Women reporting a PPBC score of 1, 2, or 3 by week 12 did not respond to therapy.
Time Frame: 12 weeks
Population: This analysis comprises women who received mirabegron and completed 12 weeks of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Mirabegron
Number analyzed (Participants) | 44
Participants
  Responded to therapy | 15
  Did not respond to therapy | 29

2. Secondary Outcome: Change in Overactive Bladder Questionnaire (OAB-q) Health Related Quality of Life (HRQL)
Description: The Overactive Bladder Questionnaire (OAB-q) Health Related Quality of Life (HRQL) score is a measure of patients' bladder symptom severity. It ranges from 25 to 150 where higher scores indicate greater quality of life.
Time Frame: 12 weeks
Population: This analysis comprises women who received mirabegron for 12 weeks and completed the Overactive Bladder Questionnaire at baseline and after 12 weeks of therapy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirabegron
Number analyzed (Participants) | 40
score on a scale
  Baseline | 50.92 (26.14)
  After 12 weeks of therapy | 74.88 (25.35)
  Change Score | 23.96 (17.54)
Statistical Analysis 1: Comparison: Mirabegron; The null hypothesis is that there is no change in patients' baseline Overactive Bladder Questionnaire (OAB-q) Health Related Quality of Life (HRQL) score after 12 weeks of therapy; Test type: Superiority; p < .0001, t-test, 2 sided; A two-sided paired t-test was used for this analysis; Mean Difference (Final Values) = 23.96, 95% CI 2-sided [18.35 to 29.57], Standard Error of Mean 2.7741

3. Secondary Outcome: Change in Urinary Distress Inventory (UDI)
Description: The Urinary Distress Inventory is a 29-item questionnaire that asks patients to report how bothered they are by symptoms of urinary urgency on a scale from 1 (not at all) to 4 (quite a bit). The total score ranges from 0 to 300 where higher scores indicate worsening symptom severity.
Time Frame: 12 weeks
Population: This analysis comprises women who received mirabegron for 12 weeks and completed the Urinary Distress Inventory at baseline and after 12 weeks of therapy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirabegron
Number analyzed (Participants) | 44
score on a scale
  Baseline | 121.25 (51.19)
  After 12 weeks of therapy | 69.62 (46.75)
  Change Score | -51.62 (40.85)
Statistical Analysis 1: Comparison: Mirabegron; The null hypothesis is that there is no change in patients' baseline Urinary Distress Inventory score after 12 weeks of therapy; Test type: Superiority; p < .0001, t-test, 2 sided; A two-sided paired t-test was used for this analysis; Mean Difference (Final Values) = -51.62, 95% CI 2-sided [-64.04 to -39.20], Standard Error of Mean 6.1584

4. Secondary Outcome: Change in Pelvic Organ Prolapse Distress Inventory (POPDI) Score
Description: The Pelvic Organ Prolapse Distress Inventory (POPDI) is a 16-item questionnaire that asks patients to report how bothered they are by symptoms of urinary urgency on a scale from 1 (not at all) to 4 (quite a bit). The total score ranges from 0 to 300 where higher scores indicate worsening symptom severity.
Time Frame: 12 weeks
Population: This analysis comprises women who received mirabegron for 12 weeks and completed the Prolapse Distress Inventory at baseline and after 12 weeks of therapy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirabegron
Number analyzed (Participants) | 44
score on a scale
  Baseline | 77.85 (64.80)
  After 12 weeks of therapy | 48.55 (50.91)
  Change Score | -29.30 (36.28)
Statistical Analysis 1: Comparison: Mirabegron; The null hypothesis is that there is no change in patients' baseline Pelvic Organ Prolapse Distress Inventory score after 12 weeks of therapy; Test type: Superiority; p < .0001, t-test, 2 sided; A two-sided paired t-test was used for this analysis; Mean Difference (Final Values) = -29.30, 95% CI 2-sided [-40.33 to -18.27], Standard Error of Mean 5.4701

5. Secondary Outcome: Change in Colo-Rectal-Anal Distress Inventory (CRADI)
Description: The Colo-Rectal-Anal Distress Inventory (CRADI) is a 17-item questionnaire that asks patients to report how bothered they are by symptoms of urinary urgency on a scale from 1 (not at all) to 4 (quite a bit). The total score ranges from 0 to 400 where higher scores indicate worsening symptom severity.
Time Frame: 12 weeks
Population: This analysis comprises women who received mirabegron for 12 weeks and completed the Colo-Rectal-Anal Distress Inventory at baseline and after 12 weeks of therapy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirabegron
Number analyzed (Participants) | 44
score on a scale
  Baseline | 94.50 (82.18)
  After 12 weeks of therapy | 62.50 (68.17)
  Change Score | -32.00 (40.61)
Statistical Analysis 1: Comparison: Mirabegron; The null hypothesis is that there is no change in patients' baseline Colo-Rectal-Anal Distress Inventory score after 12 weeks of therapy; Test type: Superiority; p < .0001, t-test, 2 sided; A two-sided paired t-test was used for this analysis; Mean Difference (Final Values) = -32.00, 95% CI 2-sided [-44.35 to -19.65], Standard Error of Mean 6.1226

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 26 weeks
Arm/Group | Mirabegron
All-Cause Mortality (participants affected / at risk) | 0/84
Serious Adverse Events (participants affected / at risk) | 2/84
Other Adverse Events (participants affected / at risk) | 12/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirabegron (N=84)
Stroke (Nervous system disorders) | 1 (1)
Breast Cancer (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirabegron (N=84)
Bacterial Infection (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Somnolence (General disorders) | 1 (1)
Leg pain (General disorders) | 1 (1)
Elevated Systolic Blood Pressure (Vascular disorders) | 2 (2)
Abdominal Cramping (Gastrointestinal disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Allergic Reaction to mirabegron (Product Issues) | 1 (1)

LIMITATIONS AND CAVEATS:
There are no limitations or caveats to report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT02495389/ICF_000.pdf
  • Study Protocol (2015-09-08): https://cdn.clinicaltrials.gov/large-docs/89/NCT02495389/Prot_001.pdf